CLINICAL TRIAL: NCT07358156
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single Dose, Phase 1 Study to Compare the Pharmacokinetics, Pharmacodynamic, Immunogenicity, and Safety of CKD-706 With US-Dupixent®, and EU-Dupixent® in Healthy Adult Participants.
Brief Title: A Study to Compare the Pharmacokinetics, Pharmacodynamic, Immunogenicity, and Safety of CKD-706 With US-Dupixent®, and EU-Dupixent® in Healthy Adult Participants.
Acronym: CKD-706
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A160_01AD2502; 2025-523115-11-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: CKD-706
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1 (Experimental): 173 healthy participants receiving one dose of investigational medical product
  Interventions: Drug: CKD-706
- Arm 2 (Active Comparator): 173 healthy participants receiving one dose of investigational medical product
  Interventions: Drug: US-Dupixent
- Arm 3 (Active Comparator): 173 healthy participants receiving one dose of investigational medical product
  Interventions: Drug: EU-Dupixent

INTERVENTIONS:
Drug: CKD-706 — One subcutaneous dose of CKD-706 in pre-filled syringe, 300 mg/2mL
  Arms: Arm 1
Drug: US-Dupixent — One subcutaneous dose of US-Dupixent in pre-filled syringe, 300 mg/2mL
  Arms: Arm 2
Drug: EU-Dupixent — One subcutaneous dose of EU-Dupixent in pre-filled syringe, 300 mg/2mL
  Arms: Arm 3

SUMMARY:
This is a randomised, double-blind, three-arm, parallel group, single-dose, Phase 1 comparative study of CKD-706, US-Dupixent, and EU-Dupixent in healthy adult participants.

DETAILED DESCRIPTION:
Dosing the CKD-706, US Dupixent, or EU-Dupixent 300 mg at Day 1. Blood samples for Pharmacokinetic analysis will be collected on Day 1 - 85. Blood sample for Pharmacodynimic and immunogenicity analysis will be collected on Day 1 - 85.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is capable of giving signed informed consent
2. Male and female healthy participant between 18 to 55 years of age (inclusive) at screening, with suitable veins for cannulation or repeated venipuncture.
3. Body-mass index between 18.5 - 29.9 kg/m2 (inclusive) with body weight ≥ 50 kg and < 95 kg at screening.
4. Participant agrees to be available for the entire duration of the study
5. All female participants must have a negative serum pregnancy test at the screening visit and on admission to the Clinical Unit (Day -1).
6. Female Participants:

   • A female participant is eligible to participate if she is not pregnant, not be lactating and not breastfeeding, and at least one of the following conditions applies
7. Male Participants • Male participants and their female spouse/partners who are of childbearing potential must be using 2 forms of birth control from screening until at least 3 months after the end of study intervention dose.

Exclusion Criteria:

1. Participant with history of any clinically important disease or disorder which, may either put the participant at risk during study.
2. Any clinically important medical/surgical procedure or trauma within 8 weeks of the screening visit, or any planned inpatient hospitalisation during the study period.
3. Participant with prior exposure to dupilumab (Dupixent or biosimilar dupilumab).
4. Participation in any interventional clinical trial or receipt of any investigational product within 30 days (or < 5 half-lives of investigational drug taken) prior to dosing.
5. Participant with current malignancy or within the past 5 years and suspected malignancy or undefined neoplasms.
6. Participant with history or presence of chronic gastrointestinal, hepatic, renal, or pancreatic disease or ongoing acute disease in these organs, or any other condition constituting a risk when taking the study intervention.
7. Participant with diagnosis or history of immunodeficiency or increased susceptibility to severe infections, or a clinically significant infection within 4 weeks of screening.
8. Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results at screening or admission, as judged by the Investigator.
9. Participant with white blood cell count < lower limit of normal at screening or admission.
10. Participant with any clinically significant abnormal finding in vital signs as judged by the Investigator.
11. Any clinically significant abnormalities on 12-lead ECG at screening or admission (Day -1) to the Clinical Unit, as judged by the Investigator.
12. Participant with positive screen results for drugs of abuse or alcohol at screening or on admission to the Clinical Unit.
13. Known or suspected history of alcohol or illicit drug abuse or excessive intake of alcohol within 1 year of screening, as judged by the Investigator.
14. Participants who smoke more than 5 cigarettes per day or consume equivalent nicotine substitutes, including e-cigarettes or inability to refrain from smoking during the in-house stay period.
15. Participant has received live vaccine(s) or live attenuated vaccines within 1 month prior to screening or plans to receive such vaccines during the study.
16. Participant with known helminthic infection, or within 6 months prior to screening.
17. Participant has a positive test for human immunodeficiency virus antibody or positive results for Hepatitis B surface antigen, anti-hepatitis B core antibody or Hepatitis C virus antibody, except for vaccinated participants or participants with past but resolved hepatitis, at screening.
18. Participant is unwilling to avoid consumption of coffee and caffeine-containing beverages within 48 hours prior to admission on Day -1 and not consuming caffeine before any outpatient visits.
19. Participant with excess use of caffeine, which is defined as exceeding 500 mg caffeine/day (e.g., > 5 cups of coffee) within 14 days prior to administration of the study intervention.
20. Participant has donated blood (> 500 mL) or blood products within 56 days prior to admission.
21. Participant has used over-the-counter medications (including vitamins), prescription medications or herbal remedies from 14 days prior to admission until the End of Study visit.
22. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to monoclonal or polyclonal antibodies. History of allergy or reaction to any formulation components of the study intervention.
23. Participant is unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope, and possible consequences of the clinical study.
24. Participant is unlikely to comply with the protocol requirements, instructions and study related restrictions.
25. Participant has previously been enrolled in this clinical study.
26. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
27. Involvement of any Chong Kun Dang Pharmaceutical, Parexel or study site employee or their close relatives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 519 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-11-16 (Estimated); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) | Day 1 - 85.
Area under the concentration-time curve from time zero up to infinity (AUC0-inf) | Day 1 - 85.
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUC0-last) | Day 1 - 85.

CONTACTS AND LOCATIONS:
Locations (2):
- Parexel EPCU Berlin, Berlin, State of Berlin, Germany
- Parexel EPCU London, London, England, United Kingdom